CLINICAL TRIAL: NCT06098209
Title: Comparing the Sedative Effect of Dexmedetomidine and Propofol in Mechanically Ventilated Patients by Using Salivary Alpha-amylase as a Stress Marker: a Randomize Controlled Trial
Brief Title: Dexmedetomidine and Propofol in Mechanically Ventilated Patients by Using Salivary Alpha-amylase as a Stress Marker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, ِAhmed Mohamed Ibrahim, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264PR353/9/23
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Dexmedetomidine; Propofol; Mechanical Ventilation; Salivary Alpha Amylase; Stress
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D (Dexmedetomidine) (Experimental): Patient will receive dexmedetomidine 0.2-1.4 μg/kg/h. Patients will be randomized to receive dexmedetomidine intravenously at rates of 0.2-1.4 μg/kg/h and 0.3-4 mg/kg/h for 2 days, respectively, to maintain the Richmond Agitation-Sedation Scale (RASS) within the range of +1 to -2.
  Interventions: Drug: Dexmedetomidine
- Group P (Propofol) (Experimental): Patient will receive propofol 0.3-4 mg/kg/h. Patients will be randomized to receive propofol intravenously at rates of 0.2-1.4 μg/kg/h and 0.3-4 mg/kg/h for 2 days, respectively, to maintain the Richmond Agitation-Sedation Scale (RASS) within the range of +1 to -2.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — Patient will receive dexmedetomidine 0.2-1.4 μg/kg/h.
  Arms: Group D (Dexmedetomidine)
Drug: Propofol — Patient will receive propofol 0.3-4 mg/kg/h.
  Arms: Group P (Propofol)

SUMMARY:
The aim of this study is to compare the efficacy of dexmedetomidine and propofol on decreasing stress in mechanically ventilated patients by using salivary alpha-amylase as a stress marker.

DETAILED DESCRIPTION:
Critically ill patients receiving mechanical ventilation (MV) in the Intensive Care Unit (ICU) have been reported to suffer due to their sense of dependency on technical medical equipment and from severe emotional responses such as hopelessness, anxiety, high levels of frustration and stress. The administration of sedatives is intended to reduce and/or prevent these negative experiences and to facilitate nursing care.

Dexmedetomidine is a highly selective α2 receptor agonist with 1600-fold affinity to α1 receptor. The use of dexmedetomidine before anesthesia has a positive effect on hemodynamic stability, which has been associated with reduced postoperative mortality and reduction of unpleasant postoperative complications . Dexmedetomidine has been shown to provide good patient comfort during MV; it also has a satisfactory safety profile and reduces time to extubating.

Salivary alpha amylase (SAA) will be considered as a suitable biomarker of sympathetic nervous system activity in recent years. SAA is locally produced by the highly differentiated epithelial acinar cells of the exocrine salivary glands, mostly of the parotid glands and plays an important role in carbohydrate hydrolysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years old.
* Both sexes.
* Newly mechanically ventilated.

Exclusion Criteria:

* Patients who used inhaled steroids.
* Patients who used any medication that could affect salivary glands (such as antihypertensive, antidepressants or antipsychotic drugs).
* Those with smoking and drinking habits.
* Patients on adrenoreceptor agonist or antagonist therapy.
* Pregnant female.
* Known hypersensitivity to the study drugs.
* Women using oral contraceptive or were in their menstrual cycle.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
The level of salivary alpha-amylase. | 2 days after intervention
  The level of salivary alpha-amylase will be measured immediately after the mechanical ventilation then after 12h for 2 days.

SECONDARY OUTCOMES:
Duration of mechanical ventilation | 28 days after intervention
  Time till weaning from mechanical ventilation
Intensive care unit length of stay | 28 days after intervention
  Time from admission till intensive care discharge
Heart rate | 2 days after intervention
  Heart rate (HR) will be recorded every 6 hours for 2 days.
Mean arterial pressure | 2 days after intervention
  Mean arterial pressure (MAP) will be recorded every 6 hours for 2 days.
Adverse events | 2 days after intervention
  Adverse events Such as hypotension and bradycardia will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.